CLINICAL TRIAL: NCT00181012
Title: Benefit of Lidocaine Perfusion in Cancer Related Visceral Pain Resistant to Morphinics: Efficacy Study in Adults and Children. Randomized Prospective Study With Direct Individual Benefit
Brief Title: Benefit of Lidocaine Perfusion in Cancer Related Visceral Pain Resistant to Morphinics
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIDODOULABDO; CSET 2003/1054
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Cancer; Pain
Keywords: Cancer Related Visceral Pain Resistant to Morphinics
MeSH Terms: conditions — Neoplasms; Pain | interventions — Lidocaine

INTERVENTIONS:
Drug: Lidocaine

SUMMARY:
This study will evaluate the benefit of lidocaine perfusion in cancer related visceral pain resistant to morphinics. It is an efficacy study in adults and children and a randomized prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from cancer of any type, at any stage, hospitalized at the Institut Gustave Roussy
* Aged from 6 to 14 years old (group A) and from 15 to 70 years old (adults)
* Presenting visceral pain due to neurotoxic chemotherapy, due to the tumoral mass or to peritoneal carcinosis
* Pain resistant to morphinic treatment

Exclusion Criteria:

* Cardiac troubles, clinical cardiac insufficiency, or history of myocardial infarction (MI) of less than 3 months
* Neurological: non-controlled epilepsy, encephalopathy, or dementia
* Severe hepatic insufficiency
* Severe renal insufficiency
* Respiratory insufficiency
* Patients having surgery or in postoperative period
* Known deficit in G6PD, alanine exposure, or sulphamide treatment
* Porphyria
* Weight > 80 kg

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-05

PRIMARY OUTCOMES:
To determine prospectively the lidocaine efficacy in 2 types of patient populations with cancer (group A: children from 6 to 14 years old and group B: adults from 15 to 70 years old) | continuous intravenous perfusion for 6 days

SECONDARY OUTCOMES:
To confirm the tolerance of the lidocaine

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Poulain, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave-Roussy, Villejuif, France